CLINICAL TRIAL: NCT02890355
Title: Randomized Phase II Study of 2nd Line FOLFIRI Versus Modified FOLFIRI With PARP Inhibitor ABT-888 (Veliparib) (NSC-737664) in Metastatic Pancreatic Cancer
Brief Title: FOLFIRI or Modified FOLFIRI and Veliparib as Second Line Therapy in Treating Patients With Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02248; NCI-2015-02248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1513; S1513 (Other: SWOG); S1513 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (veliparib and mFOLFIRI) (Experimental): Patients receive veliparib PO BID every 12 hours on days 1-7, irinotecan hydrochloride IV over 90-120 minutes on day 3, leucovorin calcium IV over 90-120 minutes on day 3, and fluorouracil IV over 46 hours on days 3-5.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Veliparib
- Arm II (FOLFIRI) (Active Comparator): Patients receive irinotecan hydrochloride IV over 90-120 minutes on day 1, leucovorin calcium IV over 90-120 minutes on day 1, and fluorouracil IV bolus over 15 minutes on days 1 and then over 46 hours on days 1-3.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Fluorouracil — Given IV bolus
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm II (FOLFIRI)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888
  Arms: Arm I (veliparib and mFOLFIRI)

SUMMARY:
This randomized phase II trial studies how well modified irinotecan hydrochloride, leucovorin calcium, fluorouracil (FOLFIRI) and veliparib as a second line of therapy work compared to FOLFIRI in treating patients with pancreatic cancer that has come back after a period of improvement (metastatic). Drugs used in chemotherapy, such as irinotecan hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether modified FOLFIRI and veliparib as second line therapy is more effective than FOLFIRI alone in treating metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall survival (OS) of metastatic pancreatic cancer patients treated with fluorouracil, irinotecan (irinotecan hydrochloride), leucovorin (leucovorin calcium), (modified FOLFIRI) and ABT-888 (veliparib) compared to a control arm of fluorouracil, irinotecan, and leucovorin (FOLFIRI).

SECONDARY OBJECTIVES:

I. To evaluate the frequency and severity of toxicity associated with each of the treatment arms in this patient population.

II. To evaluate the progression-free survival (PFS) in each of the treatment arms in this patient population.

III. To evaluate the overall response rate (confirmed and unconfirmed; complete response + partial response), disease control rate (confirmed and unconfirmed; complete response + partial response + stable disease), and duration of response in each of the treatment arms in this patient population.

TERTIARY OBJECTIVES:

I. To evaluate if breast cancer, early onset (BRCA)1 and BRCA2 mutations (somatic or germline) are associated with improved clinical outcomes (overall survival [OS], progression-free survival [PFS] and overall response rates [ORR]) in each treatment arm.

II. To evaluate the impact of homologous recombination deficiency (HRD) score on clinical outcomes in each treatment arm.

III. To evaluate the impact of genomic alterations identified by the BROCA-homologous recombinant (HR) assay, other than BRCA1/2, on clinical outcomes in each treatment arm.

IV. To bank tissue for future translational medicine studies.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive veliparib orally (PO) twice daily (BID) every 12 hours on days 1-7, irinotecan hydrochloride intravenously (IV) over 90-120 minutes on day 3, leucovorin calcium IV over 90-120 minutes on day 3, and fluorouracil IV over 46 hours on days 3-5.

ARM II: Patients receive irinotecan hydrochloride IV over 90-120 minutes on day 1, leucovorin calcium IV over 90-120 minutes on day 1, and fluorouracil IV bolus over 15 minutes on days 1 and then over 46 hours on days 1-3.

In both arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented pancreatic adenocarcinoma; patients with pancreatic neuroendocrine tumors, lymphoma of the pancreas, or ampullary cancer are not eligible
* Patients must have metastatic disease that is measurable; computed tomography (CT) scans or magnetic resonance imaging (MRI)s used to assess measurable disease must have been completed within 28 days prior to registration; CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients must not have history of brain metastases
* Patients must have had one and only one prior regimen of systemic therapy for metastatic disease unless the patient meets the criteria below
* Prior systemic therapy and chemoradiotherapy for treatment of resectable, borderline resectable or locally advanced unresectable disease is allowed and does not count toward prior therapy for metastatic disease
* Patients who received systemic therapy with gemcitabine/nab-paclitaxel for resectable or borderline/locally advanced unresectable disease and progressed with metastatic disease within 3 months of the past dose of systemic therapy are eligible
* Patients must have completed systemic therapy at least 14 days prior to registration, any surgical procedure must have been performed at least 14 days prior to registration, and radiation therapy must be completed at least 7 days prior to registration; patients must have recovered from major side effects of prior therapies or procedures in the opinion of the local site investigator prior to registration
* Patients must not have received prior irinotecan-based chemotherapy (e.g. irinotecan hydrochloride, leucovorin calcium, fluorouracil, and oxaliplatin [FOLFIRINOX] or FOLFIRI)
* Patients must not have received prior PARP inhibitor therapy including, but not limited to ABT-888, olaparib, rucaparib, and talazoparib (BMN637)
* Patients must have a Zubrod performance status of 0-1
* Within 14 days prior to registration: Absolute neutrophil count (ANC) >= 1,500/mcL
* Within 14 days prior to registration: Hemoglobin >= 9 g/dL
* Within 14 days prior to registration: Platelets >= 100,000/mcL
* Within 14 days prior to registration: Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Within 14 days prior to registration: Serum albumin >= 3.0 g/dL
* Within 14 days prior to registration: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN; patients with liver metastases may have AST and ALT of =< 5.0 x IULN
* Within 14 days prior to registration: Serum creatinine =< 2.0 mg/dL
* Patients must have CA19-9 obtained within 14 days prior to registration; if CA19-9 is normal a carcinoembryonic antigen (CEA) must be tested within 14 days prior to registration
* Patients must have blood urea nitrogen (BUN), alkaline phosphatase, sodium, potassium, calcium, glucose, chloride, and bicarbonate levels obtained within 14 days prior to registration
* Patients must not have any clinically significant and uncontrolled major medical condition(s) including, but not limited to uncontrolled nausea/vomiting/diarrhea; active uncontrolled infection; symptomatic congestive heart failure (New York Heart Association [NYHA] class >= II); unstable angina pectoris or cardiac arrhythmia; psychiatric illness/social situation that would limit compliance with study requirements
* Patients must not have active seizure or history of seizure
* Patients must be able to swallow whole capsule
* Patients must have a complete physical examination and medical history within 28 days prior to registration
* Patients must not have known Gilbert's syndrome
* Patients must not have known hypersensitivity to irinotecan, fluorouracil, or leucovorin
* Patients of childbearing potential must have a negative pregnancy test within 28 days prior to registration and must not be nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method during the study and for 6 months following completion of treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must be willing and able to undergo a biopsy after signed consent and prior to registration; patients must have tumor tissue and blood samples available and be willing to submit tumor and blood samples; NOTE: core biopsy required; fine needle aspiration (FNA) is not an acceptable substitute for core biopsy
* If archival tumor is available for submission, patients must be willing to submit tumor sample
* Patients must be offered the opportunity to participate in specimen banking for future use
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elena G Chiorean, Principal Investigator — SWOG Cancer Research Network
Locations (783):
- United States (783):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Garnet Health Medical Center, Middletown, New York
  - University of Rochester, Rochester, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was designed to enroll 143 patients, but was closed early based on the results of a planned interim futility analysis. Thus, only 123 patients were enrolled on the study.
Pre-assignment Details: 123 participants were enrolled, but 4 were ineligible and 2 refused assigned FOLFIRI treatment. Thus, 117 were eligible for analyses.
Groups:
- Arm I (Veliparib and mFOLFIRI): Participants receive veliparib PO BID every 12 hours on days 1-7, irinotecan hydrochloride IV over 90-120 minutes on day 3, leucovorin calcium IV over 90-120 minutes on day 3, and fluorouracil IV over 46 hours on days 3-5.
  Fluorouracil: Given IV
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
  Veliparib: Given PO
- Arm II (FOLFIRI): Participants receive irinotecan hydrochloride IV over 90-120 minutes on day 1, leucovorin calcium IV over 90-120 minutes on day 1, and fluorouracil IV bolus over 15 minutes on days 1 and then over 46 hours on days 1-3.
  Fluorouracil: Given IV
  Fluorouracil: Given IV bolus
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
Period: Overall Study
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Started | 59 | 58
Treated & Assessed for AEs | 56 | 50
Completed | 0 | 0
Not Completed | 59 | 58
Not completed — Adverse Event | 5 | 5
Not completed — Refusal unrelated to adverse event | 5 | 10
Not completed — Progression/relapse | 46 | 39
Not completed — Not protocol specified | 3 | 4

BASELINE CHARACTERISTICS:
Population: All eligible participants that were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI) | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Median (Full Range); unit: years] | 67 [45 to 85] | 67 [39 to 84] | 67 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 31 | 33 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 52 | 47 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Prior treatment for metastic pancreatic adenocarcinoma [Count of Participants; unit: Participants]
  Yes | 53 | 52 | 105
  No | 6 | 6 | 12
Zubrod (ECOG) Performance Status [Count of Participants; unit: Participants] — Scale: 0-5, with 0 denoting perfect health and 5 death. 0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 14 | 23 | 37
    1 | 45 | 35 | 80

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS: time to death by any cause from randomized treatment arm assignment.
  The log-rank test with stratification was used by prior systemic treatment for metastatic disease. Distributions of overall survival in arms 1 and 2 were estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Population: All eligible participants according to the intent-to-treat principle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Number analyzed (Participants) | 59 | 58
months | 5.4 [3.7 to 7.2] | 6.5 [5.6 to 7.8]
Statistical Analysis 1: Comparison: Arm I (Veliparib and mFOLFIRI) vs Arm II (FOLFIRI); Test type: Superiority; p = 0.28, Log Rank — a priori threshold for statistical significance, one sided p=0.02; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.85 to 1.78]

2. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Arm I Veliparib and mFOLFIRI: Participants receive veliparib PO BID every 12 hours on days 1-7, irinotecan hydrochloride IV over 90-120 minutes on day 3, leucovorin calcium IV over 90-120 minutes on day 3, and fluorouracil IV over 46 hours on days 3-5.
  Fluorouracil: Given IV
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
  Veliparib: Given PO
- Arm II FOLFIRI: Participants receive irinotecan hydrochloride IV over 90-120 minutes on day 1, leucovorin calcium IV over 90-120 minutes on day 1, and fluorouracil IV bolus over 15 minutes on days 1 and then over 46 hours on days 1-3.
  Fluorouracil: Given IV
  Fluorouracil: Given IV bolus
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
Arm/Group | Arm I Veliparib and mFOLFIRI | Arm II FOLFIRI
Number analyzed (Participants) | 56 | 50
Participants
  Abdominal infection | 0 | 1
  Abdominal pain | 2 | 1
  Acute coronary syndrome | 1 | 0
  Alanine aminotransferase increased | 2 | 0
  Alkaline phosphatase increased | 2 | 3
  Anemia | 4 | 5
  Anorexia | 3 | 0
  Aspartate aminotransferase increased | 1 | 1
  Atrial fibrillation | 0 | 1
  Atrial flutter | 0 | 1
  Blood bilirubin increased | 4 | 5
  Cardiac disorders - Other, specify | 1 | 0
  Catheter related infection | 1 | 0
  Confusion | 0 | 1
  Cough | 0 | 1
  Dehydration | 6 | 1
  Device related infection | 1 | 0
  Diarrhea | 6 | 3
  Dyspnea | 1 | 0
  Enterocolitis infectious | 0 | 1
  Fall | 0 | 1
  Fatigue | 10 | 3
  Febrile neutropenia | 1 | 1
  Fever | 0 | 1
  Generalized muscle weakness | 2 | 1
  Hyperglycemia | 1 | 1
  Hypertension | 1 | 2
  Hypokalemia | 2 | 1
  Hyponatremia | 2 | 3
  Hypotension | 0 | 1
  Infections and infestations - Other, specify | 2 | 1
  Lymphocyte count decreased | 3 | 6
  Mucositis oral | 0 | 1
  Nausea | 7 | 2
  Neutrophil count decreased | 20 | 11
  Platelet count decreased | 4 | 0
  Sepsis | 1 | 0
  Thromboembolic event | 1 | 0
  Vascular disorders - Other, specify | 1 | 0
  Vomiting | 5 | 2
  White blood cell decreased | 7 | 3

3. Secondary Outcome: Progression Free Survival (PFS)
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive without report of progression are censored at date of last contact.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
Population: All eligible participants according to the intent-to-treat principle.
Measure: Median (99% Confidence Interval); unit: months
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Number analyzed (Participants) | 59 | 58
months | 2.1 [1.9 to 2.4] | 2.9 [2.2 to 4.2]
Statistical Analysis 1: Comparison: Arm I (Veliparib and mFOLFIRI) vs Arm II (FOLFIRI); Test type: Superiority; p = 0.09, Log Rank; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.96 to 2.02]

4. Secondary Outcome: Overall Response Rate, ORR
Description: Overall response rate (ORR) is defined as the proportion of participants who have a confirmed and unconfirmed, partial or complete response to therapy.
Time Frame: Up to 3 years post registration
Population: Eligible participants with measurable disease.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Number analyzed (Participants) | 57 | 51
proportion of participants | 0.09 [0.01 to 0.16] | 0.10 [0.02 to 0.18]

5. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) is defined as the proportion of participants who have a confirmed and unconfirmed, partial, complete or stable response to therapy.
Time Frame: Up to 3 years post registration
Population: Eligible participants with measurable disease.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Number analyzed (Participants) | 57 | 51
proportion of participants | 0.32 [0.19 to 0.44] | 0.47 [0.33 to 0.61]

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR: time from date of first documentation of response (complete response, CR, or partial response, PR) to date of first documentation of progression or symptomatic deterioration, or death due to any cause among participants, who achieve a response (CR or PR).
  The distribution of DoR in each treatment arm will be estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years post registration
Population: Eligible participants with measurable disease, and who had confirmed partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Veliparib and mFOLFIRI) | Arm II (FOLFIRI)
Number analyzed (Participants) | 3 | 3
months | 3.4 [2.6 to 3.4] | 5.1 [2.2 to 5.2]

7. Other Pre Specified Outcome: Prevalence of BRCA1 and BRCA2 Mutations (Somatic or Germline)
Description: BRCA1/2 mutations will be associated with clinical outcomes (OS, PFS, and overall response rate [ORR]).
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Homologous Recombination Deficiency (HRD) Score
Description: The impact of HRD positivity will be evaluated on clinical outcomes in each treatment arm. The HRD score is the unweighted sum of loss of heterozygosity footprint, telomeric allelic imbalance, and large-scale state transitions measurements on a scale from 0-100. The HRD score threshold for positivity in this population will be estimated by applying receiver operating characteristic curves, classifying patients by overall disease response.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Genomic Alterations Identified by the BROCA-homologous Recombinant (HR) Assay
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. All adverse events, regardless of attribution or grade, are reported for patients who received study treatment.
  All eligible participants were assessed for All-Cause Mortality
  Only participants that received protocol treatment were assessed for Serious and Other (Not Including Serious) Adverse Events), Therefore, the 11 participants in the initial cohort that refused protocol therapy were excluded.
Arm/Group | Arm I Veliparib and mFOLFIRI | Arm II FOLFIRI
All-Cause Mortality (participants affected / at risk) | 56/59 | 56/58
Serious Adverse Events (participants affected / at risk) | 23/56 | 6/50
Other Adverse Events (participants affected / at risk) | 55/56 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Veliparib and mFOLFIRI (N=56) | Arm II FOLFIRI (N=50)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Endocrine disorders-Other (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Jejunal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 2 | 0
Fatigue (General disorders) | 3 | 0
Fever (General disorders) | 2 | 2
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 6 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
Vascular disorders-Other (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Veliparib and mFOLFIRI (N=56) | Arm II FOLFIRI (N=50)
Anemia (Blood and lymphatic system disorders) | 25 | 29
Sinus tachycardia (Cardiac disorders) | 3 | 1
Blurred vision (Eye disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 17 | 13
Ascites (Gastrointestinal disorders) | 2 | 3
Bloating (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 17 | 12
Diarrhea (Gastrointestinal disorders) | 31 | 31
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Flatulence (Gastrointestinal disorders) | 7 | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 6
Mucositis oral (Gastrointestinal disorders) | 7 | 9
Nausea (Gastrointestinal disorders) | 31 | 26
Oral pain (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 20 | 16
Chills (General disorders) | 3 | 6
Edema limbs (General disorders) | 7 | 9
Fatigue (General disorders) | 32 | 30
Fever (General disorders) | 6 | 11
Flu like symptoms (General disorders) | 3 | 2
Pain (General disorders) | 5 | 9
Infections and infestations-Other (Infections and infestations) | 4 | 4
Fall (Injury, poisoning and procedural complications) | 4 | 3
Alanine aminotransferase increased (Investigations) | 14 | 13
Alkaline phosphatase increased (Investigations) | 17 | 21
Aspartate aminotransferase increased (Investigations) | 14 | 15
Blood bilirubin increased (Investigations) | 7 | 11
Creatinine increased (Investigations) | 7 | 3
INR increased (Investigations) | 4 | 1
Investigations-Other (Investigations) | 5 | 5
Lymphocyte count decreased (Investigations) | 19 | 23
Neutrophil count decreased (Investigations) | 29 | 22
Platelet count decreased (Investigations) | 15 | 14
Weight loss (Investigations) | 15 | 9
White blood cell decreased (Investigations) | 26 | 22
Anorexia (Metabolism and nutrition disorders) | 24 | 13
Dehydration (Metabolism and nutrition disorders) | 8 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 15
Hypokalemia (Metabolism and nutrition disorders) | 12 | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 14 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6
Dizziness (Nervous system disorders) | 6 | 9
Dysgeusia (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 2 | 5
Memory impairment (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 5
Tremor (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 7 | 2
Depression (Psychiatric disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 8 | 8
Proteinuria (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 4
Hot flashes (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 8 | 6
Hypotension (Vascular disorders) | 4 | 2
Thromboembolic event (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02890355/Prot_SAP_000.pdf